CLINICAL TRIAL: NCT02058225
Title: Developing Advanced MRI Methods for Detecting the Impact of Nutrients on Infant Brain Development
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Ellen Grant, MD, Boston Children's Hospital
Other Study IDs: 84421489-1
Record Dates: First submitted 2014-02-04; First posted 2014-02-10 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Infant Development
Keywords: Infant Nutrition; Magnetic resonance spectroscopy; Infant Brain Development; Diffusion weighted Imaging; Diffusion tensor tractography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infant Group 1: This group consist of healthy, full-term babies whose mothers have no known medical conditions or complications during pregnancy.

SUMMARY:
The purpose is to study the effect of infant nutrition on brain development, as measured using Magnetic Resonance (MR) techniques. The investigators will collect detailed information about the diet of each of the infants, and seek to correlate this information with multiple MR measurements, including structural imaging, diffusion imaging, and functional connectivity. The MR scans will be performed at birth and 3 months of age. Dietary information collected will include detailed food diaries describing the feeding habits of the infants, and food frequency questionnaires to characterize the diet of the mother.

DETAILED DESCRIPTION:
The purpose is to study the effect of infant nutrition on brain development, as measured using Magnetic Resonance (MR) techniques. The investigators will collect detailed information about the diet of each of the infants, and seek to correlate this information with multiple MR measurements, including structural imaging, diffusion imaging, and functional connectivity. The MR scans will be performed at birth and 3 months of age. Dietary information collected will include detailed food diaries describing the feeding habits of the infants, and food frequency questionnaires to characterize the diet of the mother.

ELIGIBILITY:
Inclusion Criteria:

* full-term babies whose mothers have no known medical conditions or complications during pregnancy.

Exclusion Criteria:

* preterm babies
* babies whose mothers have significant medical conditions and/or significant complications during pregnancy.

Max Age: 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The participants are recruited from two major hospitals at the bedside soon after normal delivery.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2017-05-22 (Actual); Study Completion 2017-05-22 (Actual)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging to measure of brain metabolites, brain structures and brain function | Infants receive an MRI at 3 months of age
Magnetic Resonance Imaging to measure of brain metabolites, brain structures and brain function | Infants receive an MRI scan at less than 2 weeks of age

SECONDARY OUTCOMES:
Nutritional analysis of mothers diet using a food frequency questionnaire | Mothers fill out questionnaire at three months after enrollment into the study

OTHER OUTCOMES:
Mullen Early scales of Learning (MSEL) test | This test is conducted with the infants at 3 months of age prior to the month MRI scan.

CONTACTS AND LOCATIONS:
Overall Officials: P Ellen Grant, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Waltham Imaging Center: Boston Childrens Hospital, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zollei L, Iglesias JE, Ou Y, Grant PE, Fischl B. Infant FreeSurfer: An automated segmentation and surface extraction pipeline for T1-weighted neuroimaging data of infants 0-2 years. Neuroimage. 2020 Sep;218:116946. doi: 10.1016/j.neuroimage.2020.116946. Epub 2020 May 20. PMID 32442637
- [Derived] Karmacharya S, Gagoski B, Ning L, Vyas R, Cheng HH, Soul J, Newberger JW, Shenton ME, Rathi Y, Grant PE. Advanced diffusion imaging for assessing normal white matter development in neonates and characterizing aberrant development in congenital heart disease. Neuroimage Clin. 2018 May 1;19:360-373. doi: 10.1016/j.nicl.2018.04.032. eCollection 2018. PMID 30013919
- [Derived] Ferradal SL, Gagoski B, Jaimes C, Yi F, Carruthers C, Vu C, Litt JS, Larsen R, Sutton B, Grant PE, Zollei L. System-Specific Patterns of Thalamocortical Connectivity in Early Brain Development as Revealed by Structural and Functional MRI. Cereb Cortex. 2019 Mar 1;29(3):1218-1229. doi: 10.1093/cercor/bhy028. PMID 29425270